CLINICAL TRIAL: NCT06842576
Title: Transition Readiness Mobile Health Intervention: Co-Design and Pilot Study
Brief Title: Health Care Transition Readiness Short-Form Video Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Caitlin Sayegh, Medical Staff/USC Faculty, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHLA-21-00158
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Health Care Transition Readiness; Health Literacy; Self Efficacy; Emotional Wellbeing; Appointment Attendance
Keywords: mobile health; health education; transition readiness; chronic illness; adolescence; health literacy; social media; video; self efficacy; emotional wellbeing
MeSH Terms: conditions — Health Education; Chronic Disease

STUDY DESIGN:
Intervention Model Description: pilot parallel randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health education videos (Experimental): The social media intervention will consist of 7 short videos between 20-60 seconds each, filmed by a professional videographer. Videos 1) start with text asking a question or giving a title highlighting the educational topic, 2) display adolescent volunteer patient partners directly teaching self-management and transition skills, demonstrating the skills via tutorials, or presenting health education content in the style of social media trends, and 3) conclude with a written summary of take-away points. The videos will be shared to participants as a password-protected Vimeo.com playlist. If participants are more comfortable in Spanish, they will be given the option to view the videos dubbed in Spanish.
  Interventions: Behavioral: Health Education Videos
- Publicly Available Health Education Website (Active Comparator): The social media intervention will be contrasted against a control condition consisting of sharing the GotTransition.org Youth and Young Adult Resources webpage: https://gottransition.org/youth-and-young-adults/. This website is a project from The National Alliance to Advance Adolescent Health. The webpage includes videos, infographics, quizzes, and frequently asked questions. Testing the social media intervention against this existing national resource will assess whether the novel intervention is relatively more acceptable or efficacious than an active comparison. If participants are more comfortable in Spanish, a prompt will be provided to them to use the website search function to locate resources in Spanish.
  Interventions: Behavioral: GotTransition.org Website

INTERVENTIONS:
Behavioral: Health Education Videos — Participants will be prompted to explore the 7 health education videos for up to 20 minutes.
  Arms: Health education videos
Behavioral: GotTransition.org Website — Participants will be prompted to explore the Gottransition.org website for up to 20 minutes
  Arms: Publicly Available Health Education Website

SUMMARY:
The goal of this clinical trial is to assess whether social-media style short-form health education videos can increase health care transition readiness, self-efficacy, emotional well-being, health literacy, and appointment attendance, compared with publicly available health education resources in adolescents with chronic illnesses. The main question it aims to answer is:

-Hypothesize social media intervention will increase health care transition readiness, self-efficacy, emotional well-being, health literacy, and appointment attendance compared to publicly available health education website immediately post intervention and at 6 month follow up.

Participants will be randomly assigned to one of the interventions and access the intervention for 20 minutes and complete 30-60 minutes of surveys.

ELIGIBILITY:
Inclusion Criteria:

* Patients in subspecialty clinics
* Between 12 and 17 years old
* With access to an internet-connected device
* Speaking English or Spanish
* With sufficient cognitive capacity to understand the study procedures, as assessed via a teach back method.

Exclusion Criteria:

* none

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Self-reported score with a range from 1-5, on the Transition Readiness Assessment Questionnaire (TRAQ). | Immediate post-treatment and 6-month follow-up.
  The TRAQ assesses the readiness of youth and young adults to transition from pediatric to adult healthcare. It includes items related to managing medications, appointment keeping, tracking health issues, and communicating with healthcare providers.
Self-reported score ranging from 1 to 4, via the Generalized Self-Efficacy Scale (GSES). | Immediate post-treatment and 6-month follow-up.
  The GSES evaluates an individual's belief in their ability to cope with a variety of difficult demands in life. It consists of 10 items, each rated on a 4-point scale, assessing confidence in handling unexpected events and solving problems.
Self-reported score ranging from 1 to 5, via the Positive and Negative Affect Schedule for Children and Adolescents (PANAS-C). | Immediate post-treatment and 6-month follow-up.
  The PANAS-C measures positive and negative affect in children and adolescents. It includes items that assess the extent to which individuals experience various positive and negative emotions over the past few weeks.
Self-report questionnaire with a score ranging from 10 to 40, via the Health Literacy for Youth. | Immediate post-treatment and 6-month follow-up.
  The HLSAC measures subjective health literacy in youth, focusing on their ability to access, understand, and use health information to make informed decisions.
Number of appointments attended divided by the number of appointments scheduled, producing a score ranging from 0 to 100%, via medical chart abstraction. | Comparing 6 months before intervention to 6 months after intervention.
  This measure calculates the percentage of scheduled medical appointments that were attended by the patient, providing insight into adherence to treatment plans and engagement with healthcare services.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin S Sayegh, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
To protect patient confidentiality, we will not share data.

REFERENCES:
- [Background] Carrera Diaz K, Yau J, Iverson E, Cuevas R, Porter C, Morales L, Tut M, Santiago A, Ghavami S, Reich E, Sayegh CS. Human-centered design approach to building a transition readiness mHealth intervention for early adolescents. J Pediatr Psychol. 2025 Jan 1;50(1):106-114. doi: 10.1093/jpepsy/jsae066. PMID 39172486
- [Background] Bal MI, Sattoe JN, Roelofs PD, Bal R, van Staa A, Miedema HS. Exploring effectiveness and effective components of self-management interventions for young people with chronic physical conditions: A systematic review. Patient Educ Couns. 2016 Aug;99(8):1293-309. doi: 10.1016/j.pec.2016.02.012. Epub 2016 Mar 3. PMID 26954345
- [Background] Modi AC, Pai AL, Hommel KA, Hood KK, Cortina S, Hilliard ME, Guilfoyle SM, Gray WN, Drotar D. Pediatric self-management: a framework for research, practice, and policy. Pediatrics. 2012 Feb;129(2):e473-85. doi: 10.1542/peds.2011-1635. Epub 2012 Jan 4. PMID 22218838